CLINICAL TRIAL: NCT01277432
Title: A Multicentre Study to Investigate the Prevalence and Factors Associated With Depression in Chinese Patients With Type 2 Diabetes
Brief Title: Prevalence Study of Depression in Chinese Patients With Type 2 Diabetes (HK13)
Acronym: DD2
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Asia Diabetes Foundation (Other)
Responsible Party: Principal Investigator, Juliana Chan, Professor Chan, Chinese University of Hong Kong
Other Study IDs: CRE-2010-281
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes; Depression
Keywords: Diabetes; Depression
MeSH Terms: conditions — Diabetes Mellitus; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Psychiatrist interview: All patients will receive the same assessments as the 'active comparator' arm, but in addition those patients found to have positive symptoms for mild to severe depression by PHQ9 or CESD (PHQ>10 and/or CES>16) and a random sample of subjects with no or mild symptoms will also undergo a face-to-face interview by a trained clinician or psychiatrist using the following instruments:
  * MINI
  * SSI-28 (somatization)
  Interventions: Other: Psychiatrist Interview
- Depression screening: All study participants will undergo a comprehensive diabetes assessment by completing a full set of questionnaires and clinical assessments, using the JADE e-portal.
  All patients will also undergo detailed psychological and behavioral assessments using validated questionnaires.
  Several specialist questionnaires will also be conducted with all patients, including those on depression, self care and quality of life;
  1. Patient Health Questionnaire (PHQ-9)
  2. Depression Anxiety and Stress Scale (DASS-21)
  3. Diabetes Distress Scale (DDS-17)
  4. Life events questions (Inter-Heart Study)
  5. Diabetes Empowerment Scale (C-DES 20)
  6. Summary of Diabetes Self Care Activities (SDSCA-15)
  7. Euroqol-5D (EQ-5D)
  Interventions: Other: Depression screening - control

INTERVENTIONS:
Other: Psychiatrist Interview — Patients will receive a face-to-face interview by a trained clinician or psychiatrist using the following instruments:
  * MINI
  * SSI-28 (somatization)
  Groups: Psychiatrist interview
Other: Depression screening - control — All study participants will undergo;
  1. a comprehensive diabetes assessment by completing a full set of questionnaires and clinical assessments, using the JADE e-portal
  2. a detailed psychological and behavioral assessments using validated questionnaires
  3. several specialist questionnaires on depression, self care and quality of life
  Groups: Depression screening

SUMMARY:
The investigators aim to:

1. Estimate the prevalence of depression in a consecutive cohort of Chinese patients diagnosed with Type 2 Diabetes (T2D) living in areas of China with different socioeconomical affluence
2. Examine patients' awareness of the frequent coexistence of these 2 conditions
3. Analyze the associations between depression and T2D, in particularly the role of metabolic control, socioeconomical status and cognitive-psychological-behavioral factors
4. To document the predisposing, precipitating and perpetuating factors for depression and their interrelationships in Chinese type 2 diabetic patients

DETAILED DESCRIPTION:
Overall objectives of this multicentre study are to document;

1. the prevalence and diagnosis rates of depression in type 2 diabetic (T2D) patients attending 7 centres in 4 major cities in China including Hong Kong (HK), Shanghai (SH), Guangzhou (GZ) and Beijing (BJ)
2. the predisposing, precipitating and perpetuating factors for depression and their interrelationships in Chinese T2D patients

This study includes two phases. In the phase I pilot study, the investigators shall confirm and compare the validity of Patient Health Questionnaire (PHQ-9) and Clinical Epidemiological Scale for Depression (CESD) in predicting depression in Chinese T2D patients using the SCID as a gold standard. Other questionaires which measure personal and external factors, diabetes associated distress and anxiety, quality of life, mental wellness, self efficacy, health-related behavior and compliance will also be used to document possible predisposing, precipitating and perpetuating factors for depression in diabetes. These results will be used to select a set of tools which are most informative in the evaluation of depression and mental wellness in T2D patients based on their predictions for health behavior, compliance and metabolic control. A random sample of 100 T2D patients will be recruited from 3 Diabetes Centres in GZ, BJ and HK who will complete a full set of questionnaires and structured clinical assessments using a web-based electronic portal. In each of the three centres, all patients found to have positive symptoms for mild to severe depression by PHQ9 or CESD (PHQ>10 and/or CES>16) and a random sample of 20 subjects with no or mild symptoms will undergo face-to-face interview by psychiatrists using the following instruments: SCID, BDI, SSI-28 (somatization), Coping (Brief Cope 28, Chinese version).

In Phase II, the investigators shall use a subset of the most informative questionaires to document the rates of depression (diagnosed and undiagnosed) and cognitive-psychological-behavioral factors in a consecutive cohort of Chinese patients with T2D and its associations with metabolic control and psychological behavioral factors. In each of the 7 participating centres in HK, SH, BJ and GZ, 500 consecutive patients will undergo comprehensive clinical assessments for risk factors, complications and medications the JADE (Joint Asia Diabetes Evaluation) e-portal, giving a total of 3500 patients.

This survey which documents the rate of depression in T2D patients using similar methodologies will provide a comprehensive data set for exploratory analysis of the multicausality and heterogeneity of clinical presentation and risk factors in Chinese populations. Once this cohort is established and subject to availability of future funding, they can be followed up prospectively to validate and discover risk factors for new onset of depression. Apart from raising awareness, these data are essential in our design of care models and interventions to tailor the unmet needs of these patients. Data from this study will also provide insights into the effects of rapid acculturation and migration on the double burden of diabetes and depression in Chinese populations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with type 2 diabetes
2. Aged ≥25 and <75 years inclusive
3. Chinese ethnicity

Exclusion Criteria:

1. Patients with mental/physical handicap and/or difficulty in communication such as deafness, mental retardation
2. Patients with disabling diseases or reduced life expectancy such as severe heart failure, stroke, respiratory diseases, or late stages of cancer
3. Patients diagnosed with type 1 diabetes, defined as presentation with diabetic ketoacidosis or unprovoked ketosis or requirement of continuous insulin requirement within 12 months of diagnosis

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Hospitals and community centre
Sampling Method: Probability Sample
Enrollment: 3218 (Actual)
Dates: Start 2010-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Depression and psychological well-being | 1 year
  1. Depression (PHQ-9, CESD)
  2. Depression Anxiety and Stress Scale (DASS-21)
  3. Diabetes Stress Scale (DSS-17)

SECONDARY OUTCOMES:
Percentage of patients who attain 2 or more of the 'ABC' targets | 1 year
  Percentage of patients who attain 2 or more of the following 3 targets:
  1. HbA1c <7%
  2. BP <130/80 mmHg
  3. LDL cholesterol <2.6 mmol/L
Self care and Efficacy | 1 year
  1. Diabetes Empowerment Scale (C-DES)
  2. Summary of Diabetes Self Care Activities (SDSCA-15)
Quality of life | 1 year
  Using EuroQol-5D (EQ-5D) tool

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (7):
- China (6):
  - 1st Affiliated Hosp, Peking University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Shanghai Sixth People's Hospital, Shanghai
- YCK Diabetes Assessment Centre, Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- See also: Works of the Asia Diabetes Foundation — http://www.adf.org.hk